CLINICAL TRIAL: NCT04587596
Title: An Exploration of the Impact of Pain Education on GP Practice Staff: a Mixed Methods Study
Brief Title: An Exploration of the Impact of Pain Education on GP Practice Staff
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Mrs Jagjit Mankelow, Principal Investigator, Teesside University
Other Study IDs: 205/18
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Staff attitudes and beliefs; Education; GP surgery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical staff: All clinical staff employed at one surgery in Middlesbrough, UK who wish to participate
  Interventions: Other: Pain education

INTERVENTIONS:
Other: Pain education — 70 minute lecture about chronic pain and one focus group afterwards
  Other Names: Pain neurophysiology education; Therapeutic neurophysiology education

SUMMARY:
The aim of the research project is to quantify GP practice staffs' knowledge of chronic pain, their attitudes towards people with chronic pain and their management of a hypothetical patient with chronic pain, following a pain education session.

The study also seeks to explore GP practice staffs' experience of receiving the pain education, their understanding of pain following the education and if they perceive the education session has impacted upon their daily practice.

DETAILED DESCRIPTION:
Inappropriate, biomedical based views of chronic pain are commonly held by health care professionals (HCPs) and these in turn can result in patients receiving sub-optimal care out of step with current guidelines. It has been found that healthcare professionals management techniques did not reflect recognised treatment guidelines and this was associated with their biomedical view of chronic pain.

Pain education/training sessions for health care staff may be an important step towards improving patient care for chronic pain. It has been found that there was improvement in nurses' knowledge after 2 different pain education sessions delivered to nurses however there was no long term follow up. Furthermore, no studies have targeted all members of staff at a GP surgery who will interact with the patient, and thus impact upon the care they receive.

Pain Neuroscience education (PNE) is an approach to pain education which uses pain science information to shift the belief system of the receiver away from a biomedical understanding of pain to a more biopsychosocial understanding of pain.

A number of studies have shown that this education can decrease biomedical attitudes in health care students. Thus, it may be that this education could produce similar positive effects in GP practice staff that could have positive implications for the care of patients with chronic pain.

Thus this study aims to assess the impact on attitudes and beliefs of pain education upon staff at a GP surgery in Middlesbrough. Attitudes and beliefs will be assessed before and after the delivery of education. In addition participants will be invited to attend one of two focus groups to further discuss their findings or thoughts about the lecture.

ELIGIBILITY:
Inclusion Criteria

* Clinical non-NHS staff at a Middlesbrough GP Surgery.

Exclusion Criteria

* Non-clinical staff at a Middlesbrough GP surgery and staff who are not directly employed by the Surgery.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All non-NHS clinical staff at Linthorpe Surgery, principally nurses and doctors.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
HC-PAIRS | 70 minutes
  Health Care Providers Pain and Impairment Relationship Scale - assessing attitudes and beliefs towards pain using a 13 item validated questionnaire. High score is a worse outcome. Scores range from 13-91.
Revised pain neurophysiology quiz | 70 minutes
  Measures knowledge of pain physiology using a 12 point validated questionnaire. Low score is poor sign. Scores range from 0-12.
case vignette | 70 minutes
  Measures clinical practise behaviours in pain management. A validated proxy measure of clinical behaviour, MCQ weighted as appropriate or inappropriate according to current national clinical guidelines. A low score is good, and scores range from 4 to 20.
Interviews - qualitative assessment | 1 hour
  Interviews to assess perception and intended application of lecture material

CONTACTS AND LOCATIONS:
Overall Officials: J Mankelow, MSc, Principal Investigator — Teesside University
Locations (1):
- Linthorpe Surgery, Middlesbrough, United Kingdom

REFERENCES:
- [Derived] Mankelow J, Ryan CG, Green PW, Taylor PC, Martin D. An exploration of primary care healthcare professionals' understanding of pain and pain management following a brief pain science education. BMC Med Educ. 2022 Mar 28;22(1):211. doi: 10.1186/s12909-022-03265-2. PMID 35351106